CLINICAL TRIAL: NCT04786015
Title: Advancing Patient Safety for Special Populations: Active Surveillance Reporting to Identify Adverse Events Following Chiropractic Care in Older Adults
Brief Title: Active Surveillance Reporting to Identify Adverse Events Following Chiropractic Care in Older Adults
Status: Active, not recruiting | Type: Observational
Sponsor: Canadian Memorial Chiropractic College (Other)
Collaborators: Parker University (Other); Macquarie University, Australia (Other); Memorial University of Newfoundland (Other)
Responsible Party: Sponsor
Other Study IDs: 202004
Record Dates: First submitted 2020-08-10; First posted 2021-03-08 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Musculoskeletal Pain; Musculoskeletal Symptoms
Keywords: Older adult; Adverse event; Patient safety
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Active Surveillance Reporting System — A system to actively record change in symptoms older adult patients experience following a chiropractic visit.

SUMMARY:
In Canada, almost 19% of chiropractic patients are aged over 65 years. Although most of patients ≥65 years seek care for musculoskeletal conditions (such as back, neck and lower limb pain), there is inadequate prospective data on the safety of chiropractic care for these patients and the frequency of potential associated adverse events remains unknown. Our study will investigate changes in symptoms reported by older adults receiving chiropractic care, with a focus on safety.

DETAILED DESCRIPTION:
Rationale: Musculoskeletal conditions are more common and more severe in older adults than in younger adults and have a negative effect on their overall health-related quality-of-life by decreasing mobility, reducing social participation and causing substantial difficulties with activities of daily living. Canada's population is rapidly aging and the socioeconomic burden associated with these conditions will continue to escalate. Indeed, older patients (≥65 years) account for 18.8% of a chiropractor's case load. Given the high proportion of older adults as chiropractic patients, research on the safety of chiropractic care for this population is critical. Previous studies have reported adverse events (AEs) following specific chiropractic techniques or as secondary outcome measures in older adults; however, there has been no attempt to prospectively capture changes in symptoms (and specifically AEs).

Purpose: To: 1) calculate the frequency of AEs reported by older adults following chiropractic care with an active surveillance reporting system; and 2) explore patient and provider factors related to changes in symptom (e.g., new, worsening, improving) following chiropractic care.

More specifically, this study will use active surveillance reporting system to track the change in symptoms experienced by older adult patients after a chiropractic visit, in comparison to before. These symptoms can be pain, stiffness, fatigue, weakness, dizziness, nausea, etc. As active surveillances track the change in all symptoms experienced by all patients in a participating clinic, no specific condition/disease is being studied, but how the symptoms experienced by older adults seeking chiropractic care for a musculoskeletal condition (such as low back, neck, hip, should pain) change.

ELIGIBILITY:
Inclusion Criteria:

* older adults (≥65 years) seeking chiropractic care

Exclusion Criteria:

* diagnosed with cognitive decline (e.g. Alzheimer's Disease, dementia), acute infections, unable to read English and no access to email.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Canadian community-based chiropractors and their older adult patients who come to their office for chiropractic care.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2021-07-05 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Change in presenting symptoms (e.g., pain, weakness, etc.) following a chiropractic visit measured by active surveillance reporting system questionnaires | up to 7 days after chiropractic visit
  An active surveillance reporting system will be used. The questionnaires have been face-validated and used in previous studies. The active surveillance system consists on 3 questionnaires to be completed by the patients regarding their symptoms (such as pain, stiffness, weakness, etc.). First questionnaire is to be completed before a chiropractic visit. Second questionnaire is to be completed immediately after chiropractic treatment is provided. Third questionnaire is to be completed 2-7 days after the chiropractic visit. Based on the answers provided in each questionnaire, the change in symptom (i.e., if the symptom improved, got worse, or if the patient is experiencing new symptoms) can be tracked and recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Canadian Memorial Chiropractic College, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided